CLINICAL TRIAL: NCT06919536
Title: Controlled Feeding With 24 Hour Recall
Status: Completed | Type: Observational
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Shannon Galyean, Assistant Professor, Registered Dietitian Nutritionist, Texas Tech University
Other Study IDs: IRB2025-157
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Evaluate Accuracy 24 Dietary Recall
Keywords: 24 hour dietary recall; self report dietary intake; food frequency questionnaire; underreporting dietary intake; overreporting dietary intake; validity of 24 hour dietary recall; nutrition self report accuracy
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Men and women, aged 18-65, any race/ethnicity with no food allergies or aversions to test foods.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — There is no intervention, this is a observational study,

SUMMARY:
This study examines how accurately adults report their food intake using a common self-report method called the 24-hour dietary recall. While this method is widely used in nutrition research, it often leads to underreporting, especially among individuals with overweight or obesity. However, it is unclear if specific foods are more likely to be misreported.

To address this, participants will be served a controlled meal containing both simple foods (e.g., fruit snacks, saltine crackers, cookies, and a coke soft drink) and mixed dishes (e.g., chicken salad, macaroni and cheese with peas). Each food item will be precisely weighed before and after consumption. The following day, participants will complete an online 24-hour recall, and the process will be repeated one week later.

The study will compare reported intake to actual intake to assess accuracy and determine whether underreporting is more common for mixed dishes. It will also explore whether reporting accuracy is influenced by body weight, gender, or race. Findings from this research may improve the understanding of self-report limitations and support the development of more accurate dietary assessment tools.

DETAILED DESCRIPTION:
This prospective observational cohort study with repeated measures investigates the accuracy of self-reported dietary intake using the 24-hour dietary recall method, specifically the Automated Self-Administered 24-hour Dietary Assessment Tool (ASA-24). Research has consistently shown that individuals underreport energy intake using self-report tools, particularly those with overweight or obesity. However, there is limited understanding of which types of foods are most prone to misreporting and whether such tendencies are consistent across time or demographic groups.

To address these gaps, this study uses a controlled feeding protocol in which participants consume a standardized lunch consisting of two mixed dishes (chicken salad and macaroni and cheese with peas) and single-item foods (e.g., fruit snacks, saltine crackers, cookies, and a coke soft drink). All foods are weighed precisely before and after consumption to the nearest 0.01g. The following day, participants complete an online 24-hour dietary recall using ASA-24. This process is repeated one week later to assess reproducibility of reporting patterns.

The primary outcome is the portion-size reporting difference between actual and reported intake for each food item. Secondary outcomes include whether mixed dishes are more inaccurately reported than discrete foods, and whether underreporting is consistent across both sessions. Additional analyses will evaluate whether underreporting varies by BMI category, gender, or race.

Participants (N=65) are adults aged 18-65 recruited from the Texas Tech University community using flyers, email announcements, and word of mouth. Inclusion criteria include availability to attend lunch visits and complete online recalls. Exclusion criteria include food allergies or aversions to the test meal.

ELIGIBILITY:
Inclusion Criteria:

* Able to attend the test site for a meal at least two times.

Exclusion Criteria:

* Any aversions to the test meal (including allergies)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will include anyone eligible based on the inclusion and exclusion criteria. Those who are 18-65 years of age are eligible, there are no other restrictions.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Per-item Portion-Size Difference (Weighed - 24-hour recall) | From enrollment to 2 weeks (1 measurement with a ASA-24 the next day, and another identical measurement with recall the next day)
  The primary outcome is the difference between the calories of weighed actual intake and the reported intake from the ASA_24

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Nutrition and Metabolic Health Initiative, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Heymsfield SB, Darby PC, Muhlheim LS, Gallagher D, Wolper C, Allison DB. The calorie: myth, measurement, and reality. Am J Clin Nutr. 1995 Nov;62(5 Suppl):1034S-1041S. doi: 10.1093/ajcn/62.5.1034S. PMID 7484918
- [Background] Foster E, Lee C, Imamura F, Hollidge SE, Westgate KL, Venables MC, Poliakov I, Rowland MK, Osadchiy T, Bradley JC, Simpson EL, Adamson AJ, Olivier P, Wareham N, Forouhi NG, Brage S. Validity and reliability of an online self-report 24-h dietary recall method (Intake24): a doubly labelled water study and repeated-measures analysis. J Nutr Sci. 2019 Aug 30;8:e29. doi: 10.1017/jns.2019.20. eCollection 2019. PMID 31501691
- [Background] Schoeller DA, Thomas D, Archer E, Heymsfield SB, Blair SN, Goran MI, Hill JO, Atkinson RL, Corkey BE, Foreyt J, Dhurandhar NV, Kral JG, Hall KD, Hansen BC, Heitmann BL, Ravussin E, Allison DB. Self-report-based estimates of energy intake offer an inadequate basis for scientific conclusions. Am J Clin Nutr. 2013 Jun;97(6):1413-5. doi: 10.3945/ajcn.113.062125. No abstract available. PMID 23689494
- [Background] Lin WY, Dubuisson O, Rubicz R, Liu N, Allison DB, Curran JE, Comuzzie AG, Blangero J, Leach CT, Goring H, Dhurandhar NV. Response to Comment on: Lin et al. Long-term changes in adiposity and glycemic control are associated with past adenovirus infection. Diabetes Care 2013;36:701-707. Diabetes Care. 2013 Sep;36(9):e162. doi: 10.2337/dc13-0879. No abstract available. PMID 23970733
- [Result] Subar AF, Crafts J, Zimmerman TP, Wilson M, Mittl B, Islam NG, McNutt S, Potischman N, Buday R, Hull SG, Baranowski T, Guenther PM, Willis G, Tapia R, Thompson FE. Assessment of the accuracy of portion size reports using computer-based food photographs aids in the development of an automated self-administered 24-hour recall. J Am Diet Assoc. 2010 Jan;110(1):55-64. doi: 10.1016/j.jada.2009.10.007. PMID 20102828
- [Result] Freedman LS, Commins JM, Moler JE, Arab L, Baer DJ, Kipnis V, Midthune D, Moshfegh AJ, Neuhouser ML, Prentice RL, Schatzkin A, Spiegelman D, Subar AF, Tinker LF, Willett W. Pooled results from 5 validation studies of dietary self-report instruments using recovery biomarkers for energy and protein intake. Am J Epidemiol. 2014 Jul 15;180(2):172-88. doi: 10.1093/aje/kwu116. Epub 2014 Jun 10. PMID 24918187
- [Result] Ahluwalia N, Dwyer J, Terry A, Moshfegh A, Johnson C. Update on NHANES Dietary Data: Focus on Collection, Release, Analytical Considerations, and Uses to Inform Public Policy. Adv Nutr. 2016 Jan 15;7(1):121-34. doi: 10.3945/an.115.009258. Print 2016 Jan. PMID 26773020